CLINICAL TRIAL: NCT06685055
Title: Identification of Clinical, Biological, Cellular and Genetic Markers of Favorable Response to Therapy With Neonatal Fc Receptor Inhibitors for Immunoglobulins (FcRn) in Patients With Generalized Myasthenia Gravis (INFORM)
Brief Title: Markers of Favorable Response to FcRn Inhibitors(INFORM)
Acronym: INFORM
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6717
Record Dates: First submitted 2024-07-10; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-07

CONDITIONS: Myasthenia Gravis Generalized
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Myasthenia gravis is an autoimmune neurological disease caused by autoantibodies primarily directed against components of the postsynaptic membrane of the neuromuscular junction. Approximately 85% of patients have antibodies directed against the acetylcholine receptor (anti-AChR).

Anti-AChR antibodies act through three distinct mechanisms:

1. Activation of the classical complement pathway: Formation of membrane-attack complexes (MACs) results in the destruction of the postsynaptic membrane.
2. Mechanical blockade: Anti-AChR antibodies block the acetylcholine binding site on its receptor.
3. Internalization and lysosomal degradation: Bivalent IgG causes cross-linking of adjacent receptors leading to internalization and degradation of AChRs (antigenic modulation).

Patient mortality has significantly reduced due to effective treatments preventing severe exacerbations of myasthenic symptoms.

In the past five years, the FDA and EMA have approved complement inhibitors and FcRn inhibitors for treating generalized myasthenia gravis with anti-AChR antibodies. Many other therapies are currently in phase 3 clinical trials or under regulatory review. However, there is no specific evidence to support which patients benefit most from one treatment class over another.

Given their relative efficacy compared to conventional therapies and high costs, their future role in the therapeutic arsenal is unclear. A personalized approach considering the different pathogenic mechanisms of anti-AChR and single gene polymorphisms involved in treatment response is essential for effective therapeutic choice. In July 2023, AIFA approved the reimbursement of Efgartigimod in Italy for treating adult patients with generalized myasthenia gravis with anti-AChR antibodies, in addition to standard therapy.

FcRn inhibitors (including Efgartigimod) prevent the interaction of IgG with the neonatal Fc receptor for immunoglobulin fragments, reducing IgG recycling and promoting the degradation of IgG and pathogenic antibodies without affecting albumin levels.

There is heterogeneity among patients in their response to FcRn inhibitors therapies. Currently, there is no specific evidence indicating which patients may benefit most from this class of treatments. Interindividual heterogeneity in the autoantibody repertoire, predominance of different pathogenic mechanisms, and single gene polymorphisms affecting treatment response. Investigating the immune profile and specific gene polymorphisms in myasthenic patients needing these innovative therapies could identify predictive biomarkers and personalize therapeutic choices.

ELIGIBILITY:
Inclusion Criteria:

- Age ≥18 years.

* Diagnosis of generalized anti-AChR positive Myasthenia Gravis.
* Need for therapy with neonatal Fc receptor inhibitors for immunoglobulins (FcRn) as per AIFA-approved therapeutic indications (14).
* Ability to follow up at the reference center.
* Signed informed consent for the study.

Exclusion Criteria:

* Age <18 years.

  * Poor compliance with drug therapy.
  * Concurrent autoimmune diseases.
  * Insufficient availability of clinical information.
  * Ongoing neoplasm or infection at the time of biological sample collection.
  * Refusal to sign the informed consent for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with generalized Myasthenia Gravis positive for anti-AChR antibodies undergoing therapy with FcRn inhibitor drugs
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2026-07-09 (Estimated); Study Completion 2026-07-09 (Estimated)

PRIMARY OUTCOMES:
Identification of Clinical Markers of Favorable Response to FcRn Inhibitors Therapy in Patients With Generalized Myasthenia Gravis | 24 months
  Analyze the clinical status of patients comparing the results of MG-ADL clinical scale pre/post FcRn Inhibitors
Identification of Biological and Cellular Markers of Favorable Response to FcRn Inhibitors Therapy in Patients With Generalized Myasthenia Gravis | 24 months
  Analyze the differences between IgG levels pre/post therapy with FcRn inhibitors
Identification of Biological and Cellular Markers of Favorable Response to FcRn Inhibitors Therapy in Patients With Generalized Myasthenia Gravis | 24 months
  • Evaluate anti-AChR positivity in patients treated with FcRn inhibitors
Identification of Biological and Cellular Markers of Favorable Response to FcRn Inhibitors Therapy in Patients With Generalized Myasthenia Gravis | 24 months
  • Dosage of proteins involved in pathogenesis
Identification of Genetic Markers of Favorable Response to FcRn Inhibitors Therapy in Patients With Generalized Myasthenia Gravis | 24 months
  Investigate the presence of polymorphisms in the FCGRT gene (VTNRs) in patients refractory to therapy with FcRn inhibitors
Identification of Clinical Markers of Favorable Response to FcRn Inhibitors Therapy in Patients With Generalized Myasthenia Gravis | 24 months
  Analyze the clinical status of patients comparing the results of QMG clinical scale pre/post FcRn Inhibitors

SECONDARY OUTCOMES:
Predictive algorithm of favorable response | 24 months
  Create a predictive algorithm for response to FcRn inhibitor therapies by combining clinical, cellular, biological, and genetic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Iorio, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy